CLINICAL TRIAL: NCT04626960
Title: ADRB3, ROCK2 and GEF Levels in Overactive Bladder Patients
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Elif Fırat, Principal Investigator, Medical Biochemistry Specialist, Pamukkale University
Other Study IDs: 2019HZDP009
Record Dates: First submitted 2020-11-02; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Overactive Bladder
Keywords: ADRB3; Biomarkers; GEF; Overactive bladder; ROCK2.
MeSH Terms: conditions — Urinary Bladder, Overactive; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: OAB patients
- Control: Healthy

SUMMARY:
Aims: To evaluate changes in levels of ADRB3, ROCK2, and GEF which have key roles in the adrenergic and cholinergic pathways of contraction-relaxation harmony in voiding physiology, and to investigate the diagnostic potential of these proteins in OAB.

Methods: This study included 60 idiopathic OAB patients and a healthy control group. All patients completed a validated OAB-V8 questionnaire. Serum levels of ADRB3, ROCK2, and GEF were examined by ELISA. ROC curves were generated to evaluate the diagnostic performance of these protein levels for OAB diagnosis.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is defined by The Standardization Subcommittee of the International Continence Society (ICS) as a symptom syndrome consisting of urgency, with or without urge incontinence, usually with frequency and nocturia, in the absence of proven infection or other obvious pathology. OAB is a clinical diagnosis and its assessment is very important, especially for evaluation of treatment effectiveness. OAB is diagnosed by symptoms only, and symptoms are subjective definitions that vary from person to person. Therefore, various scoring systems and urodynamic tests are used to make an objective diagnosis and to determine the severity of symptoms. In recent studies, there are several substances that have been proposed as biomarkers of OAB, such as especially urinary proteins but studies that have compared these markers are lacking, also these proteins present low sensitivity and specificity. In the future, physicians may consider the use of biomarkers to identify distinct OAB phenotypes, with distinct causal mechanisms, selecting patients for specific target therapies with expected better outcomes. Biomarkers can be useful to phenotype patients and for selecting more effective target therapies. So, there is a need for stable and non-invasive biomarkers that can be used reliably for assessment of OAB.

Even though the exact cause or causes of OAB have not yet been identified, the most powerful theory accepted in pathogenesis is detrusor muscle hyperactivity by relaxation decrease or contractions increase in detrusor smooth muscle. The molecular mechanisms underlying the OAB clinic are still not fully understood.

Bladder contractions are primarily controlled by parasympathetic cholinergic pathways. Guanine nucleotide exchange factors (GEF) and Rho-related kinase (ROCK) are important in this way. ROCKs are also important regulators of cellular apoptosis, growth, metabolism, and migration through control of the cell contraction. GEFs activate small GTPases and they are regulatory factors that facilitate the separation of GDP from Rho and the binding of GTP. GEF protein regulates Rho activity. Overexpression of GEF leads to an increase in GTP-dependent Rho. GTP-dependent Rho enables ROCK2 activation. ROCK2 especially has an important role in regulating smooth muscle contraction. So, functional disorder or alteration in levels of GEF and ROCK2 can cause an excessive contraction in smooth muscle and may be effective in the basis of pathophysiology in OAB.

The relaxation of the bladder smooth muscle is controlled by a sympathetic cholinergic pathway in which adrenergic receptor β3 (ADRB3) plays a major role. They have an important role in regulating smooth muscle tone, especially in the bladder, and show their effect in many tissues, such as adipose tissue, through relaxation or thermogenesis. The hypofunction of this receptor causes disruption of the bladder detrusor muscle and dysfunction of the urinary tract. So a decrease in ADRB3 levels may be responsible for reduced relaxation in the pathophysiology of overactive bladder.

The aim of this study was to understand whether ADRB3, ROCK2, and GEF levels could be auxiliary parameters for the evaluation of the molecular mechanisms of OAB and to diagnose. If changes in levels of these parameters affect the amounts and functions of proteins in these pathways, the pathogenesis of OAB can be better understood and new treatment goals can be recommended.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Idiopathic Overactive Bladder
* Must have at least 11 points on the OAB-V8 questionnaire

Exclusion Criteria:

* Neurogenic bladder
* Bladder obstruction
* Urinary tract diseases such as stones, tumors, infections
* Long QT syndrome
* Severe liver failure
* Renal failure
* Myasthenia
* Glaucoma
* Autoimmune disease
* Lower urinary tract dysfunction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult OAB patients and healthy controls
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-06-07 (Actual)

PRIMARY OUTCOMES:
Serum ADRB3 levels | 2019
  Measurement of serum ADRB3 levels
Serum GEF levels | 2019
  Measurement of serum GEF levels
Serum ROCK2 levels | 2019
  Measurement of serum ROCK2 levels

CONTACTS AND LOCATIONS:
Overall Officials: Elif Fırat, Principal Investigator — elifbasak43@hotmail.com; Hülya Aybek, Study Chair — haybek@pau.edu.tr; Zafer Aybek, Study Director — zaybek@pau.edu.tr
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Meng E, Lin WY, Lee WC, Chuang YC. Pathophysiology of Overactive Bladder. Low Urin Tract Symptoms. 2012 Mar;4 Suppl 1:48-55. doi: 10.1111/j.1757-5672.2011.00122.x. PMID 26676700
- [Background] Antunes-Lopes T, Cruz F. Urinary Biomarkers in Overactive Bladder: Revisiting the Evidence in 2019. Eur Urol Focus. 2019 May;5(3):329-336. doi: 10.1016/j.euf.2019.06.006. Epub 2019 Jun 21. PMID 31231010